CLINICAL TRIAL: NCT05770479
Title: Assessing and Improving the Durability of Compensatory Cognitive Training for Older Veterans (AID-CCT)
Brief Title: Assessing and Improving the Durability of Compensatory Cognitive Training for Older Veterans
Acronym: AID-CCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E3821-W; 1IK2RX003821-01A1 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-03-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognitive Rehabilitation; Cognitive Training; Cognitive Remediation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ME-CCT Booster Training (Experimental): 3-4 Sessions of ME-CCT Booster Training
  Interventions: Behavioral: Motivationally-Enhanced Compensatory Cognitive Training (ME-CCT) Booster Modules
- Treatment as Usual (Other): Treatment as Usual
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Motivationally-Enhanced Compensatory Cognitive Training (ME-CCT) Booster Modules — ME-CCT is a traditionally a manualized group-based behavioral intervention (8 weeks, 2 hours per week) designed to improve cognitive and everyday functioning in patients with MCI. Our booster modules will be shortened and distilled from ME-CCT using the IM Adapt protocol (and thus will not be new information but rather 'reminder' content) for a personalized four-session sequence of booster training targeted toward specific everyday functional needs of individual participants.
  Other Names: ME-CCT Booster
  Arms: ME-CCT Booster Training
Other: Treatment As Usual — Treatment for MCI is generally managed by Primary Care or Neurology. Participants will continue to receive their usual care with their current providers. With no effective pharmacological treatment known for persons with MCI, providers tend to focus on encouraging a healthy lifestyle, prevention and management of modifiable risk factors for cognitive impairment, and treatment of behavioral and psychiatric symptoms.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
Veterans have numerous risk factors (e.g., PTSD, TBI, cerebrovascular problems) for later-life cognitive and functional decline. Evidence supports the effectiveness of strategy-based cognitive rehabilitation therapies, including compensatory cognitive training (CCT), for such decline. However, questions remain about the length of time that CCT-driven improvements in cognitive and everyday function last, and whether additional 'booster' training sessions could provide additional benefit to aging Veterans who previously underwent treatment. This study examines the long-term durability of CCT in Veterans aged 55+ and provides an opportunity to develop and pilot test a series of CCT booster sessions that can be personalized toward individual everyday functional goals.

DETAILED DESCRIPTION:
The RCT portion of this study is a pilot trial evaluating the feasibility and acceptability of a "booster" CCT intervention for individuals who have already previously participated in CCT. 28 Veterans who previously participated in the ME-CCT intervention group of the "Cognitive Rehabilitation for Older Veterans with Mild Cognitive Impairment" study [PI: Twamley, VA CSRD: I01CX001592] will be recruited to participate in this pilot RCT.

All participants will receive an initial assessment that consists of neuropsychological and functional capacity tests, and will complete several self-reports of quality of life and daily function. Participants will complete questionnaires focused on acceptability, appropriateness, and feasibility. Participants will then be randomized to pilot RCT booster training or Treatment as Usual (TAU) group, yielding approximately 14 participants in each group. Participants will receive either three to four booster intervention modules/sessions or treatment as usual. Directly following the approximately 4-week intervention window, all 28 participants will receive the same battery of tests and questionnaires they received at the beginning of the sub-study.

Although the investigators will attempt to estimate possible initial effects of the CCT booster on cognitive and functional outcomes, the purpose of this pilot RCT is to examine feasibility and acceptability, not to complete an adequately-powered efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 55 and older who are able to provide informed consent
* Previous completion of the "Cognitive Rehabilitation for Older Veterans with Mild Cognitive Impairment" [PI: Twamley, VA CSRD: I01CX001592] study and received the ME-CCT intervention
* Independently living
* English-speaking: this is necessary to complete cognitive and functional testing and participate in booster development and other study procedures

Exclusion Criteria:

* Participation in sub-study 2 of this CDA, in which study participants assist with the design of booster intervention modules
* DSM-5 criteria for current substance use disorder and has been substance abstinent for less than 30 days
* History of schizophrenia, schizoaffective disorder, or other primary psychotic disorder
* History of significant brain injury with loss of consciousness >30 minutes
* Auditory or visual impairments that would prevent ability to participate in booster sessions or ability to benefit from compensatory strategies

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
"Acceptability of Intervention Measure (AIM)" questionnaire mean score | 4 weeks
  Four-item measure of perceived intervention implementation acceptability from Weiner et al., (2017) that has demonstrated strong psychometric properties. On a scale of 1-5 (completely disagree to completely agree), participants are asked to respond to the following: 1) implementation strategy meets my approval 2) implementation strategy is appealing to me 3) I like the implementation strategy 4) I welcome the implementation strategy. Average score of these four questions is calculated for measure score. Mean of participants' measure scores will be reported.
"Intervention Appropriateness Measure (IAM)" questionnaire mean score | 4 weeks
  Four-item measure of perceived intervention implementation appropriateness from Weiner et al., (2017) that has demonstrated strong psychometric properties. On a scale of 1-5 (completely disagree to completely agree), participants are asked to respond to the following: 1) implementation strategy seems fitting 2) implementation strategy seems suitable 3) implementation strategy seems applicable 4) implementation strategy seems like a good match. Average score of these four questions is calculated for measure score. Mean of participants' measure scores will be reported.
"Feasibility of Intervention Measure (FIM)" questionnaire mean score | 4 weeks
  Four-item measure of perceived intervention implementation feasibility from Weiner et al., (2017) that has demonstrated strong psychometric properties. On a scale of 1-5 (completely disagree to completely agree), participants are asked to respond to the following: 1) implementation strategy seems implementable 2) implementation strategy seems possible 3) implementation strategy seems doable 4) implementation strategy seems easy to use. Average score of these four questions is calculated for measure score. Mean of participants' measure scores will be reported.

SECONDARY OUTCOMES:
Initial estimate of change in objective cognitive performance composite z score | baseline, 4 weeks
  Change in composite z score
Initial estimate of change in functional capacity performance composite z score | baseline, 4 weeks
  Change in composite z score

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline E Maye, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No